CLINICAL TRIAL: NCT00003903
Title: An Evaluation of the Effect of Androgen Ablation on Bone Resorption in Prostate Cancer Patients
Brief Title: Effect of Androgen Suppression on Bone Loss in Patients With or Without Bone Metastases Secondary to Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: CDR0000067078; P30CA011198 (NIH); URCC-U2898; NCI-G99-1522
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Osteoporosis; Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; osteoporosis
MeSH Terms: conditions — Osteoporosis; Prostatic Neoplasms

INTERVENTIONS:
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Assessing the effect of androgen suppression on bone loss in prostate cancer patients may improve the ability to plan treatment, may decrease the risk of fractures and bony pain, and may help patients live more comfortably.

PURPOSE: Clinical trial to determine the effect of androgen suppression on bone loss in patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the effect of androgen ablation on bone resorption in patients with or without bone metastases secondary to prostate cancer.

OUTLINE: Patients are stratified according to prior androgen ablation therapy (yes vs no) and metastatic disease (yes vs no).

Patients undergo blood work and 24 hour urine collection on day 1 and at week 6-8. Patients who have received androgen ablation therapy and are found to have increased bone resorption undergo a dual energy x-ray absorptiometry (DEXA) scan.

A comparison is made between androgen ablation therapy and bone resorption and if metastases are associated with the two.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer
* Stratum 1 (androgen ablation therapy):

  * Bone metastases
  * Prior orchiectomy allowed
  * Prior or concurrent leuprolide and/or goserelin therapy allowed
* Stratum 2 (androgen ablation therapy):

  * No bone metastases
  * Prior orchiectomy allowed
  * Prior or concurrent leuprolide and/or goserelin therapy allowed
* Stratum 3 (no androgen ablation therapy):

  * No metastatic disease
  * Prior flutamide or bicalutamide therapy allowed

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Calcium normal

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* See Disease Characteristics
* No concurrent high dose steroids

Radiotherapy:

* Prior radiotherapy allowed

Surgery:

* See Disease Characteristics
* Prior radical prostatectomy allowed

Other:

* No concurrent bisphosphonates

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 1999-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak M. Sahasrabudhe, MD, Study Chair — James P. Wilmot Cancer Center
Locations (1):
- James P. Wilmot Cancer Center, Rochester, New York, United States